CLINICAL TRIAL: NCT05189730
Title: Selected Chemotherapy Combined Immunotherapy Treated High Risk Patient After Neoadjuvant Chemoradiotherapy in Resected Locally Advanced Esophageal Squamous Cell Carcinoma: an Exploratory Study
Brief Title: Selected Chemotherapy Combined Immunotherapy Treated High Risk Patient After NCRT in Resected Locally Advanced ESCC
Acronym: ETNT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yongtao Han, Chief of Thoracic Surgery, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCCH-TS2107
Record Dates: First submitted 2021-11-26; First posted 2022-01-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: neoadjuvant treatment; immunotherapy; chemoradiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total neoadjuvant therapy (Experimental): The patients would receive neoadjuvant chemoradiotherapy treatment firstly. And then evaluated efficacy according to RECIST 1.1. If patients with cCR would receive surgery treatment after 4-6 weeks. After surgery, patients with pCR would always perform surveillance and patients with non-pCR would receive immunotherapy alone treatment. If patients evaluated as PD, they would receive new treatment regimen after MDT discussed. Other patients with PR and SD would receive 2 cycles of neoadjuvant immunochemotherapy. And then, Efficacy of immunochemotherapy would be evaluated according to RECIST 1.1. For patients suitable for surgery, surgery should be performed after 4-6 weeks of immunotherapy. After surgery, the patients with R0 resection would divided into two groups, if patients with pCR would always perform surveillance and patients with non-pCR would receive immunotherapy treatment. Other patients without R0 resection would receive new treatment regimen after MDT discussed.
  Interventions: Drug: Tirelizumab; Drug: Paclitaxel; Drug: Carboplatin; Radiation: Neoadiuvant radiotherapy

INTERVENTIONS:
Drug: Tirelizumab — Two cycles of Tirelizumab (200mg administered as an intravenous infusion over 30 minutes per 3 weeks), D1.
Drug: Paclitaxel — Two cycles of paclitaxel (135mg/m2 administered as an intravenous infusion per 3 weeks), D1.
Drug: Carboplatin — Two cycles of carboplatin(AUC=5 administered as an intravenous infusion per 3 weeks) D1.
Radiation: Neoadiuvant radiotherapy — Simultaneous radiotherapy would be consecutively performed for 4 weeks with the total dose of 40Gy (40Gy/ 4W /20F), D1.

SUMMARY:
Tislelizumab combined with chemotherapy sequential neoadjuvant therapy for non-cCR patients after neoadjuvant chemoradiotherapy in locally advanced ESCC. And then the patients would receive surgery and adjuvant therapy according to the postoperative pathological results. It is expected that through this study, some high-risk patients could obtain better efficacy and prolong patient survival. At same time, low risk patients could avoid increasing perioperative complications and surgical risks, so that more patients could benefit from neoadjuvant treatment. The investigators aimed to explore a more accurate comprehensive treatment mode for patients with esophageal squamous cell carcinoma, and provide a certain scientific basis for the formulation of esophageal cancer diagnosis and treatment norms in China.

ELIGIBILITY:
Inclusion Criteria:

* 1.Histologically confirmed ESCC；
* 2.Clinical stage T2N0-1M0, T3N0M0, T3N1M0, T1-3N2M0（II-III) (AJCC 8 TNM classif tion);
* 3.Locally advanced ESCC that can be treated surgically evaluated before treatment;
* 4.At least one measurable lesion in accordance with RECIST 1.1;
* 5.Have a performance status of 0 or 1 on the ECOG Performance Scale;
* 6.Expected survival time is greater than 6 months;
* 7.The important organs functions meet the following requirements:the absolute neutrophil count(ANC) ≥1.5×109/L; the platelet count ≥100×109/L; hemoglobin ≥90g/L; bilirubin is less than or equal to 1.5 times ULN, ALT and AST less than or equal 2.5 times UILN; creatinine clearance rate(CCr) ≥50mL/min; the thyroid function is normal;
* 8.Female subjects of childbearing potential have a negative pregnancy test and must agree to take effective contraceptive measures during the study period and within 3 months after the last dose;
* 9.Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

* 1.The patient have received radiotherapy, chemotherapy, hormone therapy, surgery, or molecular-targeted therapy;
* 2.Confirmed patients with distant metastasis by CT imaging;
* 3.The subject has previous or co-existing other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* 4.The subject had previously received other anti-pd-1 antibody therapy or other immunotherapy targeting pd-1 / pd-L1;
* 5.Patients with active autoimmune disease or documented autoimmune disease or symptoms requiring systemic hormone therapy or anti-autoimmune drug therapy;
* 6.Patients with immunodeficiency or who were still receiving systemic steroid hormone therapy (prednisone > 10 mg/ day or other equivalent drugs) or other forms of immunosuppressive therapy 7 days prior to the first dose of neoadjuvant therapy in this study;
* 7.Clinical ascites or pleural effusion requiring therapeutic puncture or drainage;
* 8.The subject with uncontrol cardiac clinical symptoms or diseases, such as :(1) nyha class 2 or more heart failure (2) unstable angina pectoris (3) myocardial infarction within 1 year (4) clinically significant ventricular or ventricular arrhythmias requiring treatment or intervention;
* 9.Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg> 2G /L), bleeding tendency or receiving thrombolytic or anticoagulant treatment;
* 10.The subject is present (within 3 months) with esophageal varices, active gastric and duodenal ulcers, ulcerative colitis, portal hypertension and other gastrointestinal diseases, or with active bleeding from unresected tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by the investigator;
* 11.Past or present severe bleeding (bleeding >30 ml within 3 months), hemoptysis (fresh blood >5 ml within 4 weeks) or thromboembolism events (including stroke events and/or TRANSIENT ischemic attack) within 12 months;
* 12.Patients with active infection who still required systemic treatment 7 days before the first dose of neoadjuvant therapy in this study;
* 13.Patients with past or present objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, severely impaired lung function, etc;
* 14.Senior or uncontrolled virus injection: HIV, TP, hepatitis virus;
* 15.Senior or uncontrolled virus injection: HIV, TP, hepatitis virus;
* 16.Patients who had participated in clinical trials of other drugs within 4 weeks;
* 17.The live vaccine was administered less than 4 weeks prior to study administration or possibly during the study period;
* 18.Have a history of mental illness or psychiatric substance abuse;
* 19.The subject cannot or does not agree to bear the cost of the self-paid portion of the examination and treatment, except for the clinical study drug, combined chemoradiotherapy, and SAE associated with the clinical study drug;
* 20.Other patients whom the medical practitioner considers inappropriate for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response rate | 3 months
  Definition of complete pathologic response is "no cancer cell, including lympho nodes" which corresponds with tumor regression score 0. Definition of pathologic response is as follows. Tumor regression score Grade 0 and 1 will be defined as "responder" and 2 and 3 will be considered as "non-responders"
Incidence of adverse events | 6 months
  Number of participants with treatment-related adverse events as assessed by Number of participants with treatment-related adverse events as assessed by treatment-related adverse events assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Clinical Complete Remission | 3 months
  The clinical complete remission rate (cCR) was defined as the proportion of patients with clinically confirmed cT0 or cN0(AJCC Cancer Staging Manual,8th ed. 2017 edition ).
Major Pathological Remission rate | 3 months
  The residual tumor after neoadjuvant treatment ≤ 10% residual tumor lesion in surgical specimen compared to baseline。
Objective Remission Rate | 3 months
  Objective response rate as assessed by RECISIST1.1 criteria, the percentage of subjects with CR or PR in the total number of subjects in the analysis data set during the period from the beginning of the treatment regimen to the disease progression date.
Rate of R0 resection | 3 months
  Measure the rate of R0 resection with all margins microscopically clear.
Events Free Survival | Through study completion, an average of 1 year.
  Event-free survival was defined as the time from the date of randomization to the date of the first documented non-fatal event (worsening cardiac function, hospitalization for congestive heart failure, liver function impairment, liver cirrhosis, transformation to AML, as defined in the protocol), or death, whichever occurred first. Participants who did not experience a non-fatal event as of the time of data cut-off (end of study), as well as participants who did not experience a non-fatal event and stopped study participation before the data cut-off, were censored as specified in the protocol.
Overall Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  Overall survival was the duration from the start of study treatment to death

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China

REFERENCES:
- [Derived] He W, Wang C, Wu L, Wan G, Li B, Han Y, Li H, Leng X, Du K, Chen H, Wang Q, Peng L. Tislelizumab Plus Chemotherapy Sequential Neoadjuvant Therapy for Non-cCR Patients After Neoadjuvant Chemoradiotherapy in Locally Advanced Esophageal Squamous Cell Carcinoma (ETNT): An Exploratory Study. Front Immunol. 2022 Jun 2;13:853922. doi: 10.3389/fimmu.2022.853922. eCollection 2022. PMID 35720312